CLINICAL TRIAL: NCT06350617
Title: Safety and Efficacy of Personalized Repetitive Transcranial Magnetic Stimulation Protocol Based on Functional Reserve to Enhance Ambulatory Function in Patients With Parkinson Disease
Brief Title: Personalized rTMS Protocol Based on Functional Reserve to Enhance Ambulatory Function in PD Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: National Research Foundation of Korea (Other); Ministry of Food and Drug Safety, Korea (Other Government); Seoul National University Hospital (Other); Bucheon St. Mary's Hospital (Other); Saint Vincent's Hospital, Korea (Other); Severance Hospital (Other); Kumoh National Institute of Technology (Unknown); NEUROPHET (Industry)
Responsible Party: Principal Investigator, Won Hyuk Chang, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-12-028
Record Dates: First submitted 2024-02-27; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Parkinson's Disease and Parkinsonism
Keywords: Parkinson's Disease; rTMS; Functional reserve
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders

STUDY DESIGN:
Intervention Model Description: prospective, single-blind with blind observer, parallel-group design, multi-center, randomized controlled clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participants, assessors, and investigators will be blinded, not be aware of the group allocation. Statistical analysis will also be conducted by data analysts without awareness of the group allocation. Only clinicians applying rTMS intervention will not be blinded, as they will apply rTMS over different stimulation sites based on the protocols. Blinding will be continued until the end of the study, including data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Ipsilateral High-Frequency (Experimental): Patients with motor priority confirmed by TUG and TUG-Cog tests.
  High-frequency (HF) rTMS over more affected primary motor cortex (M1) of lower extremity will be applied.
  Interventions: Device: High-Frequency, ipsilateral M1
- Bilateral High-Frequency1 (Active Comparator): Patients with motor priority confirmed by TUG and TUG-Cog tests.
  High-frequency (HF) rTMS over bilateral M1 of lower extremities will be applied.
  Interventions: Device: High-Frequency, bilateral M1
- DLPFC High-Frequency (Experimental): Patients with cognitive priority confirmed by TUG and TUG-Cog tests.
  High-frequency (HF) rTMS over Lt. dorsolateral prefrontal cortex (DLPFC) will be applied.
  Interventions: Device: High-Frequency, Lt. DLPFC
- Bilateral High-Frequency2 (Active Comparator): Patients with cognitive priority confirmed by TUG and TUG-Cog tests.
  High-frequency (HF) rTMS over bilateral M1 of lower extremities will be applied.
  Interventions: Device: High-Frequency, bilateral M1

INTERVENTIONS:
Device: High-Frequency, ipsilateral M1 — rTMS intervention: 20 sessions of 10-Hz rTMS at 90% resting motor threshold (RMT), 50 pulses per session with a 25-second interval between sessions, totaling 1,000 pulses.
  rTMS target: ipsilateral primary motor cortex of lower extremity.
  Total rTMS sessions: once a day, 5 days per 2 weeks, for 4 weeks, totaling 10 sessions.
  Additional treatment: Treadmill gait training after the intervention, as well as the routine pharmacotherapy based on the guidelines for management of patients with Parkinson's disease.
  Arms: Ipsilateral High-Frequency
Device: High-Frequency, bilateral M1 — rTMS intervention: 20 sessions of 10-Hz rTMS at 90% resting motor threshold (RMT), 50 pulses per session with a 25-second interval between sessions, totaling 1,000 pulses.
  rTMS target: bilateral primary motor cortex of lower extremity.
  Total rTMS sessions: once a day, 5 days per 2 weeks, for 4 weeks, totaling 10 sessions.
  Additional treatment: Treadmill gait training after the intervention, as well as the routine pharmacotherapy based on the guidelines for management of patients with Parkinson's disease.
  Arms: Bilateral High-Frequency1
Device: High-Frequency, Lt. DLPFC — rTMS intervention: 20 sessions of 10-Hz rTMS at 90% resting motor threshold (RMT), 50 pulses per session with a 25-second interval between sessions, totaling 1,000 pulses.
  rTMS target: Lt. DLPFC
  Total rTMS sessions: once a day, 5 days per 2 weeks, for 4 weeks, totaling 10 sessions.
  Additional treatment: Treadmill gait training after the intervention, as well as the routine pharmacotherapy based on the guidelines for management of patients with Parkinson's disease.
  Arms: DLPFC High-Frequency
Device: High-Frequency, bilateral M1 — rTMS intervention: 20 sessions of 10-Hz rTMS at 90% resting motor threshold (RMT), 50 pulses per session with a 25-second interval between sessions, totaling 1,000 pulses.
  rTMS target: bilateral primary motor cortex of lower extremity.
  Total rTMS sessions: once a day, 5 days per 2 weeks, for 4 weeks, totaling 10 sessions.
  Additional treatment: Treadmill gait training after the intervention, as well as the routine pharmacotherapy based on the guidelines for management of patients with Parkinson's disease.
  Arms: Bilateral High-Frequency2

SUMMARY:
The objective of this study was to determine the effects of protocols of repetitive transcranial magnetic stimulation (rTMS) therapy based on the functional reserve of each patient with Parkinson's disease, compared to conventional high-frequency rTMS therapy on bilateral primary motor cortex (M1). Investigators hypothesized that the functional reserve of each patient with Parkinson's disease will be different, and therefore an appropriate simulating target for rTMS therapy is needed. In addition, this approach could be more effective compared to conventional protocols applied to patient with Parkinson's disease regardless of their severity, predicted mechanism of motor function recovery, or functional reserves.

DETAILED DESCRIPTION:
rTMS treatment for patients with Parkinson's disease is traditionally based on stimulating the neural network of brain. The widely-used traditional rTMS treatment protocol involves high-frequency stimulation over the bilateral primary motor cortex (M1) to enhance motor and gait functions. However, concerns have arisen regarding the effect of rTMS on motor recovery in patients with Parkinson's disease. Although still subject to debate, a possible reason for the diverse results of rTMS applied is the uniform application protocol to individuals with varying pathologies and functional reserves, aimed at enhancing recovery.

Therefore, this study was aimed to determine the effects of protocols of rTMS therapy based on the functional reserve of each patient with Parkinson's disease.

Based on screening evaluations (Timed Up and Go Test (TUG), Timed Up and Go Dual Task-Cognitive (TUG-Cog)), investigators hypothesized that patients could be categorized into two groups: 1) priority in motor functional reserve, 2) priority in cognitive functional reserve. For each group, investigators plan to randomly assign patients to experimental and control groups to demonstrate the efficacy of different rTMS protocols based on functional reserves compared to conventional high-frequency rTMS applied to the bilateral M1.

ELIGIBILITY:
Inclusion Criteria:

1. patients with Parkinson's disease, diagnosed by the United Kingdom (UK) Parkinson's Disease Society Brain Bank Diagnostic Criteria,
2. Modified Hoehn and Yahr (H&Y) scale, stage 2~4,
3. patients who can walk on flat surfaces without the need for a gait aid,
4. aged ≥50 years old,
5. patients willing to sign the informed consent.

Exclusion Criteria:

1. those with contraindications to rTMS, such as epilepsy, implanted metal objects in the head, or a history of craniotomy,
2. those with cognitive impairment, confirmed through the Montreal Cognitive Assessment (MoCA) test as follows: < 7 points: Illiterate < 13 points: Education duration 0.5-3 years < 16 points: Education duration 4-6 years < 19 points: Education duration 7-9 years < 20 points: Education duration 10 years or more
3. those with coexisting neurological conditions, such as spinal cord injury or Stroke,
4. those with major psychiatric disorders, such as major depression, schizophrenia, or dementia,
5. those with severe on-off phenomena or severe dyskinesia, deemed by the investigators to render participation in the study inappropriate.
6. those having contraindications to conduct an MRI study,
7. those who are pregnant or lactating,
8. patients who have refused to participate in this study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Differences of Timed Up and Go Test (TUG) | From baseline T0 to Post-intervention T2 (4 weeks)
  Measurement for gait function.

SECONDARY OUTCOMES:
Differences of Timed Up and Go Test (TUG) | From baseline T0 to During-intervention T1 (2 weeks)
  Measurement for gait function.
Differences of Timed Up and Go Test (TUG) | From baseline T0 to Follow-up T3 (2 months)
  Measurement for gait function.
Differences of Timed Up and Go Test-Cognitive (TUG-Cog) | From baseline T0 to During-intervention T1 (2 weeks)
  Measurement for gait and cognitive function.
Differences of Timed Up and Go Test-Cognitive (TUG-Cog) | From baseline T0 to Post-intervention T2 (4 weeks)
  Measurement for gait and cognitive function.
Differences of Timed Up and Go Test-Cognitive (TUG-Cog) | From baseline T0 to Follow-up T3 (2 months)
  Measurement for gait and cognitive function.
Differences of Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS), Part III | From baseline T0 to Post-intervention T2 (4 weeks)
  Measurement for motor function of patients with Parkinson's disease. Score ranges from 0 to 132; higher score indicates more severity of disease status
Differences of MDS-UPDRS, Part III | From baseline T0 to Follow-up T3 (2 months)
  Measurement for motor function of patients with Parkinson's disease. Score ranges from 0 to 132; higher score indicates more severity of disease status
Differences of New Freezing of Gait Questionnaire (FoG-Q) | From baseline T0 to Post-intervention T2 (4 weeks)
  Measurement for gait function of patients with Parkinson's disease Score ranges from 0 to 28; higher score indicates more severity of disease status
Differences of New Freezing of Gait Questionnaire (FoG-Q) | From baseline T0 to Follow-up T3 (2 months)
  Measurement for gait function of patients with Parkinson's disease Score ranges from 0 to 28; higher score indicates more severity of disease status
Differences of Digit span Test | From baseline T0 to Post-intervention T2 (4 weeks)
  Measurement for cognitive function
Differences of Digit span Test | From baseline T0 to Follow-up T3 (2 months)
  Measurement for cognitive function
Differences of Trail making Test | From baseline T0 to Post-intervention T2 (4 weeks)
  Measurement for cognitive function
Differences of Trail making Test | From baseline T0 to Follow-up T3 (2 months)
  Measurement for cognitive function
Differences of Gait lab parameter (Gait speed) | From baseline T0 to Post-intervention T2 (4 weeks)
  Measurement for gait function. Gait speed (km/hr) will be measured
Differences of Gait lab parameter (Gait speed) | From baseline T0 to Follow-up T3 (2 months)
  Measurement for gait function. unit: km/hr Gait speed (km/hr) will be measured
Differences of Gait lab parameter (Stride length) | From baseline T0 to Post-intervention T2 (4 weeks)
  Measurement for gait function Stride length (m) will be measured
Differences of Gait lab parameter (Stride length) | From baseline T0 to Follow-up T3 (2 months)
  Measurement for gait function Stride length (m) will be measured
Differences of Gait lab parameter (Step count) | From baseline T0 to Post-intervention T2 (4 weeks)
  Measurement for gait function Step count will be measured
Differences of Gait lab parameter (Step count) | From baseline T0 to Follow-up T3 (2 months)
  Measurement for gait function Step count will be measured
Differences of Gait lab parameter (Cadence) | From baseline T0 to Post-intervention T2 (4 weeks)
  Measurement for gait function Cadence (step count/min) will be measured
Differences of Gait lab parameter (Cadence) | From baseline T0 to Follow-up T3 (2 months)
  Measurement for gait function Cadence (step count/min) will be measured
Differences of Gait lab parameter (Swing ratio) | From baseline T0 to Post-intervention T2 (4 weeks)
  Measurement for gait function Swing ratio (% of swing phase of 1 gait cycle) will be measured
Differences of Gait lab parameter (Swing ratio) | From baseline T0 to Follow-up T3 (2 months)
  Measurement for gait function Swing ratio (% of swing phase of 1 gait cycle) will be measured
Differences of Gait lab parameter (Stride time) | From baseline T0 to Post-intervention T2 (4 weeks)
  Measurement for gait function Stride time (unit- second, time from heel strike to next heel strike) will be measured
Differences of Gait lab parameter (Stride time) | From baseline T0 to Follow-up T3 (2 months)
  Measurement for gait function Stride time (unit- second, time from heel strike to next heel strike) will be measured
Differences of Gait lab parameter (Pressure distribution) | From baseline T0 to Post-intervention T2 (4 weeks)
  Measurement for gait function Pressure distribution (unit - pecentage, pressure distribution among heel, mild, and toe) will be measured
Differences of Gait lab parameter (Pressure distribution) | From baseline T0 to Follow-up T3 (2 months)
  Measurement for gait function Pressure distribution (unit - pecentage, pressure distribution among heel, mild, and toe) will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Won Hyuk Chang, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yun SJ, Lee HS, Kim DH, Im S, Yoo YJ, Kim NY, Lee J, Kim D, Park HY, Yoon MJ, Kim YS, Chang WH, Seo HG. Efficacy of personalized repetitive transcranial magnetic stimulation based on functional reserve to enhance ambulatory function in patients with Parkinson's disease: study protocol for a randomized controlled trial. Trials. 2024 Aug 16;25(1):543. doi: 10.1186/s13063-024-08385-2. PMID 39152467